CLINICAL TRIAL: NCT05970302
Title: XELOX and Bevacizumab in Combination With Tislelizumab for First-Line Treatment of Patients With MSS/pMMR RAS-mutated Metastatic Colorectal Cancer (mCRC): A Single-arm, Phase II Study.
Brief Title: XELOX +Bev +Tislelizumab for First-line Treatment of MSS/pMMR RAS-mutated mCRC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, LIN YANG, chief physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC-009591
Record Dates: First submitted 2023-07-06; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Tislelizumab; Bevacizumab; Oxaliplatin; Capecitabine; MSS/pMMR; Metastatic Colorectal Cancer (mCRC); RAS-mutated; First-Line
Keywords: Single-arm; Phase II
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XELOX +Bev +Tislelizumab (Experimental): Every 3 weeks as a cycle:
  1. Tislelizumab: 200mg, iv, d1;
  2. Bevacizumab: 7.5mg/kg, iv, d1;
  3. Oxaliplatin: 130mg/m2, iv, d1;
  4. Capecitabine: 1000mg/m2, bid, po, d1-d14; Re-evaluate patients every two cycles. If the patient has been treated for more than 8 cycles, they will enter maintenance therapy, and the regimen is capecitabine + BEV combined with tislelizumab.
  Interventions: Drug: Tislelizumab+Bevacizumab+Oxaliplatin+Capecitabine

INTERVENTIONS:
Drug: Tislelizumab+Bevacizumab+Oxaliplatin+Capecitabine — Use the above medications on a regular basis.

SUMMARY:
The goal of this clinical trial is to compare XELOX +Bev +Tislelizumab with standard chemotherapy，in MSS/pMMR-type RAS-mutated metastatic colorectal adenocarcinoma. The main questions it aims to answer are efficacy and safety of the regimen of XELOX +Bev +Tislelizumab. The investigators want to transform ras-mutated colorectal cancer into a "hot tumor" through the combination of anti-vascular therapy and chemotherapy, and then achieve better therapeutic effect through the combination with immunotherapy. Participants will receive the regimen of XELOX +Bev +Tislelizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed initially unresectable MSS/pMMR-type RAS-mutant metastatic colorectal adenocarcinoma;
2. ECOG score of 0 or 1;
3. Ability to swallow oral medications;
4. Have at least one measurable lesion (according to RECIST v1.1 standard);
5. No anti-tumor treatment has been received after recurrence and metastasis;
6. Neoadjuvant or adjuvant chemotherapy containing fluorouracil drugs is allowed before or after radical resection of colorectal cancer, but the treatment needs to be completed for ≥ 6 months; if oxaliplatin is used in neoadjuvant or adjuvant chemotherapy, it includes The oxaliplatin regimen needs to be completed for ≥12 months;
7. Adequate organ function: On the premise of no component blood transfusion within 14 days: white blood cells ≥ 3.5*10^9/L and neutrophils ≥ 1.5*10^9/L, hemoglobin ≥ 90g/L, platelets ≥ 100* 10^9/L; serum bilirubin ≤ 1.5 times the normal value, alanine aminotransferase (ALT) ≤ 2.5 times the normal value, aspartate aminotransferase (AST) ≤ 2.5 times the normal value; Urinary protein <2+. Or urine protein 2+ but 24-hour urine protein quantity ≤ 1 g; serum creatinine ≤ 1.5 times of normal value, creatinine clearance rate ≥ 60ml/min; Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥ lower limit of normal value (50%);
8. Expected survival period ≥ 3 months;
9. Patients fully understand this research, voluntarily participate in this clinical trial and sign an informed consent;
10. Women with reproductive potential (< 2 years after the last menstrual period) and men use effective contraceptive methods until half a year after the last treatment.

Exclusion Criteria:

1. Previously received bevacizumab or anti-CTLA4, anti-PD-1/PD-L1 therapeutic antibodies or pathway-targeted drugs;
2. Received radiotherapy within 4 weeks before the evaluation;
3. Symptomatic peripheral neuropathy > grade 2 (CTCAE5.0 standard);
4. Received live vaccine or systemic immune stimulant (including but not limited to interferon or interleukin 2) within 1 month;
5. HIV-positive and other immunodeficiency diseases;
6. Active hepatitis B or hepatitis C (except for those who have been infected or cured before, that is, HBsAg negative and hepatitis B core antigen anti-HBc antibody positive; except for hepatitis C patients whose HCV RNA is negative by PCR);
7. Existing autoimmune diseases or other diseases that require immunosuppressant treatment, except for type 1 diabetes; except for hypothyroidism that only requires hormone replacement therapy; skin diseases that do not require systemic treatment (such as vitiligo, psoriasis, alopecia areata); inhaled or topical steroids or equivalent steroids in excess of 10 mg prednisone per day, except for inactive autoimmune disease on adrenal replacement therapy;
8. Received systemic hormone therapy or treatment with a daily dose of more than 10 mg prednisone equivalent dose or other forms of immunosuppressive treatment within 7 days, but inhaled or topical steroids or daily application of more than 10 mg prednisone, etc. Except for inactive autoimmune diseases treated with adrenal replacement therapy with potent steroids;
9. Have a history of organ transplantation;
10. Uncontrolled central nervous system (CNC) metastasis (symptomatic or metastatic sites are midbrain, pons, medulla or spinal cord) or other central nervous system diseases;
11. Those who have undergone major surgery, open biopsy or obvious traumatic trauma within 1 month, or who may need major surgery during the study period; those who have undergone open biopsy or obvious traumatic trauma, or may need major surgery during the study period;
12. Combined with other malignant tumors other than intestinal cancer (except cured basal cell carcinoma or squamous cell carcinoma of the skin and carcinoma in situ of the cervix; the treatment of other malignant tumors has been completed for more than 1 year, and there is no clinical and imaging evidence of recurrence or progression except);
13. Combined active and refractory infection;
14. Cardiovascular diseases with clinical significance, such as cardiovascular accident (CVA) (≤ 6 months before treatment), myocardial infarction (≤ 6 months before treatment), unstable angina, chronic heart failure of NYHA ≥ 2 (CHF), uncontrolled arrhythmia; uncontrolled hypertension; thromboembolic or bleeding events within 6 months before treatment;
15. Evidence of causing coagulation disease;
16. With dysphagia, active peptic ulcer, complete or incomplete intestinal obstruction, active gastrointestinal bleeding, perforation, malabsorption syndrome or uncontrollable gastrointestinal inflammatory disease (such as Crohn's disease or ulcerative colon inflammation);
17. Severe unhealed wounds/ulcers or severe fractures;
18. Any serious acute or chronic medical condition that may affect the patient's participation in the study or interfere with the interpretation of the study results;
19. There are mental illnesses, serious social and psychological illnesses, or researchers believe that there are factors that may affect research compliance;
20. Pregnant or lactating women;
21. No therapeutic anticoagulant or antiplatelet drugs or NSAIDs (aspirin ≤ 325 mg/day allowed);
22. Severe allergic reaction to the test drug;
23. Reluctance to use alternative therapies such as (but not limited to) bisphosphonates if receiving RANKL inhibitors (eg, denosumab).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  ORR of regimen of XELOX +Bev +Tislelizumab

SECONDARY OUTCOMES:
Duration of Response (DoR) | 2 years
Disease Control Rate (DCR); | 2 years
Median Progression-Free Survival (mPFS) | 2 years
12-month PFS rate | 12 months
Median Overall Survival (mOS) | 5 years
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 2 years
  Adverse Events (AEs) Incidence, Serious Adverse Events (SAE) Incidence

CONTACTS AND LOCATIONS:
Locations (1):
- Lin Yang, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided